CLINICAL TRIAL: NCT01325831
Title: Change of Dopamine Pathway After rTMS Treatment in Major Depressive Disorder
Brief Title: Changes of Functional Connectivity After rTMS in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2008-0525
Record Dates: First submitted 2009-07-07; First posted 2011-03-30 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcranial magnetic stimluation (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)
- rTMS_sham (Sham Comparator)
  Interventions: Device: Sham repetitive transcranial magnetic stimulation(rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation(rTMS) — 10-day course of 10 Hz rTMS on left dorsolateral prefrontal cortex of the subjects.
  Other Names: MAGSTIM
  Arms: transcranial magnetic stimluation
Device: Sham repetitive transcranial magnetic stimulation(rTMS) — Sham repetitive transcranial magnetic stimulation(rTMS)
  Arms: rTMS_sham

SUMMARY:
In order to explore the effect of repetitive TMS, which has shown to be effective in intractable depression, we will examine resting-state, default-mode network functional connectivity in patients with major depression. We will use a double-blind, sham-controlled design. Our target sample size is 60(30 patients will be treated by active rTMS, the other 30 will be treated by sham rTMS). We will apply 10-day course of 10 Hz rTMS on left dorsolateral prefrontal cortex of the subjects.

DETAILED DESCRIPTION:
Up to now, 24 patients with major depression and 6 normal controls are enrolled. Twenty-three patients and 4 normal participants have taken 10 days rTMS. One patients and one control withdrew their consent without any reason and one control withdrew the consent because of headache.

We scanned fMRIs(to examine functional connectivity)twice for each participant, which were taken 3 days before the first and 3 days after the last rTMS.

All of participants have not reported side effects except mild headahe. There's been no seizure event up to now.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV major depressive episode
* Failure of at least 3 different kind of antidepressant

Exclusion Criteria:

* Organic brain disorder
* Other diagnosis of DMS-IV except nicotine dependence
* History of seizure disorder

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change of functional connectivity between pre/post rTMS | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: EUN LEE, M.D., Ph.D., Principal Investigator — Yonsei University College of Medicine, Severance Hospital
Locations (1):
- Department of Psychiatry, Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang JI, Lee H, Jhung K, Kim KR, An SK, Yoon KJ, Kim SI, Namkoong K, Lee E. Frontostriatal Connectivity Changes in Major Depressive Disorder After Repetitive Transcranial Magnetic Stimulation: A Randomized Sham-Controlled Study. J Clin Psychiatry. 2016 Sep;77(9):e1137-e1143. doi: 10.4088/JCP.15m10110. PMID 27379563